CLINICAL TRIAL: NCT03853213
Title: Investigating Fear Of Recurrence as a Modifiable Mechanism of Behavior Change to Improve Medication Adherence in Acute Coronary Syndrome Patients
Brief Title: Investigating Fear Of Recurrence as a Modifiable Mechanism of Behavior Change
Acronym: INFORM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Jeffrey Birk, Instructor in Medical Sciences, Columbia University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: AAAR9458; R21HL145970-01 (NIH)
Record Dates: First submitted 2019-02-22; First posted 2019-02-25 (Actual); Results first posted 2021-07-26 (Actual); Last update posted 2021-09-17 (Actual); Status verified 2021-08

CONDITIONS: Acute Coronary Syndrome; Fear; Medication Adherence
Keywords: Fear of Recurrence; Acute Coronary Syndrome; Intervention; Cognitive Bias Modification Training; Attentional Bias; Interpretation Bias; Medication Adherence
MeSH Terms: conditions — Acute Coronary Syndrome; Medication Adherence

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitive Bias Modification Training (Experimental): Participants in this intervention group complete two tasks, each repeated 8 times over the course of 4 weeks (twice per week). The first task is Cognitive Bias Modification Training for Attention. It is designed to reinforce attention away from ACS threat-related stimuli (e.g., "death," "chest pain") and toward neutral stimuli (e.g., "curve," barn doors"). The second task is Cognitive Bias Modification Training for Interpretation. It is designed to train participants to appraise ambiguous information that is potentially related to ACS threat as benign.
  Interventions: Behavioral: Cognitive Bias Modification Training
- Attention Control Training (Sham Comparator): Participants in this placebo control group complete two tasks, each repeated 8 times over the course of 4 weeks (twice per week). The first task is the placebo version of Cognitive Bias Modification Training for Attention. It is designed NOT to train attention toward or away from threatening or neutral information. The second task is the placebo version of Cognitive Bias Modification Training for Interpretation. It is designed NOT to train the interpretation of information as either threatening or benign.
  Interventions: Behavioral: Attention Control Training

INTERVENTIONS:
Behavioral: Cognitive Bias Modification Training — In task 1, participants view a pair of threat-neutral words and then a single letter (E or F). Participants' task is to tap a button as quickly and accurately as possible to indicate whether they see E or F. The letter appears in the neutral location on 90.6% of trials, thereby reinforcing participants' attending away from threat. In task 2, participants view a word or phrase corresponding to a threatening (e.g., "dying") or benign (e.g., "sleep") interpretation of a sentence (e.g., "You have been waking up tired recently"). They are asked to tap a button to indicate whether the word or phrase was related to the sentence. Positive feedback ("Correct") is given for rejected threat interpretations and for benign interpretations. Otherwise, negative feedback ("Incorrect") is given.
  Other Names: Cognitive-Affective Fear of Recurrence Intervention
  Arms: Cognitive Bias Modification Training
Behavioral: Attention Control Training — In task 1, participants view a pair of threat-neutral words and then a single letter (E or F). Participants' task is to tap a button as quickly and accurately as possible to indicate whether they see E or F. The target letter is equally likely to appear in the threat location as the neutral location. Thus, participants' patterns of attention are not trained toward or away from threat. In task 2, participants view a word or short phrase corresponding to either a threatening or benign interpretation of a sentence that follows it. They are asked to tap a button to indicate whether the word or phrase was related to the sentence. Positive feedback and negative feedback are equally likely to be given regardless of whether participants endorse the threatening or benign interpretations.
  Arms: Attention Control Training

SUMMARY:
The primary goal of this project is to identify, measure, and influence fear of cardiac event recurrence, a candidate mechanism of change in medication adherence in patients with suspected acute coronary syndrome (ACS). An intervention will be tested that has been used to reduce fear of cancer recurrence by changing emotion-related patterns of attention allocation and interpretation of neutral stimuli. Secondarily, the study will test whether a reduction in fear of cardiac event recurrence improves medication adherence.

DETAILED DESCRIPTION:
Acute coronary syndrome (ACS; myocardial infarction or unstable angina) is a leading cause of morbidity and mortality in the U.S., with >1 million cases per year. Survivors are at high risk for recurrent cardiovascular disease (CVD) events, particularly if they do not adhere to risk-reducing medications. Unfortunately, nonadherence among ACS patients is very common (~50%), and no effective, scalable interventions exist. Addressing medication nonadherence in ACS patients requires an experimental medicine approach to identify specific mechanisms of behavior change in populations for whom those mechanisms are most relevant and modifiable.

Accumulating evidence suggests that the many patients who develop post-traumatic stress disorder (PTSD) symptoms following ACS view their medications as reminders of their cardiac event and their future CVD risk. Ironically, although it has rarely been studied outside of cancer survivors, this fear of recurrence (FoR) may undermine medication adherence in ACS patients. This project will use the Science of Behavior Change (SOBC) experimental medicine approach to investigate FoR as a putative mechanism of behavior change with respect to heart medication adherence among ACS patients with early PTSD symptoms at hospital discharge. The study will test a cognitive-affective intervention that has been shown to reduce FoR in cancer survivors, that is delivered electronically (electronic tablet) in the patient's home. The intervention has been adapted in this study for ACS to be tested using a double-blind randomized controlled design. One hundred suspected ACS patients will be enrolled who reported at least mild to moderate threat perceptions at the time of their initial visit to the emergency department. FoR and future time perspective will be assessed within six weeks of the initial visit to the emergency department, and then participants will be trained on the tablet intervention. Participants will complete the intervention over four weeks in eight half-hour sessions, twice each week. Medication adherence will be measured electronically using eCAP devices. FoR and future time perspective will be reassessed 1 month after the baseline session, and cognitive-affective change will be assessed electronically throughout the intervention period.

In addition to investigating FoR as the primary mechanism of behavior change, the study also investigates a secondary potential mechanism that is a distinct, but related, construct: future time perspective. Furthermore, in addition to examining medication adherence as the primary health behavior of interest, the study also examines a secondary health behavior that is reduced in fearful cardiac patients: physical activity. Collectively, the three aims below address these two putative mechanisms (FoR, future time perspective) and these two health behaviors (medication adherence, physical activity) in the randomly assigned groups (intervention, control).

Objectives

Aim 1 (main purpose of the trial):

The study will determine whether a tablet-based cognitive bias modification treatment (CBMT) intervention influences the two putative mechanisms of fear of recurrence (FoR) and future time perspective. Of primary importance within this first aim, it will test whether the intervention reduces cardiac-related FoR relative to control. The trial is statistically powered to test the first aim as it relates to FoR. Secondarily, it will also test whether the intervention increases an expansive future time perspective relative to control.

Aim 2 (exploratory):

The study will determine the extent to which the two potential mechanisms of behavior change-FoR and future time perspective-are each associated with health behaviors. Of primary importance within this second aim, it will test associations between these two potential mechanisms of behavior change and objectively measured and self-reported adherence to heart medications (antiplatelets to reduce risk of blood clotting, antihypertensive drugs to reduce blood pressure, or statins to lower cholesterol). Of secondary importance, it will test whether these two potential mechanisms of behavior change are associated with self-reported physical activity.

Aim 3 (exploratory):

The study will test whether the intervention improves the two health behaviors of interest. Of primary importance within this third aim, it will test whether the intervention relative to control is associated with higher heart medication adherence (objectively measured or self-reported) in the two months after the baseline visit and whether any such beneficial effects are mediated by reductions in the putative mechanisms of FoR or future time perspective. Secondarily, it will test whether the intervention relative to control is associated with greater increases in self-reported physical activity in the two months after the baseline visit and whether any such beneficial effects are mediated by reductions in the putative mechanisms of FoR or future time perspective.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older;
2. Fluent in English or Spanish;
3. A diagnosis of NSTEMI or unstable angina (UA) according to American College of Cardiology criteria;
4. Currently enrolled in the protocol titled "Testing biopsychosocial mechanisms of the posthospital syndrome [PHS] model of early rehospitalization in cardiac patients" (IRB-AAAR7350 at CUIMC)
5. Previously indicated "YES" to the following question in the consent form for the separate protocol (IRB-AAAR7350) in which they are enrolled and willing to be contacted about other future research projects.
6. Elevated Threat Perception score in emergency department flagged by automatic scoring (i.e., ≥ 10, the median for 1,000 ACS patients in a separate sample)
7. Currently on a daily aspirin regimen prescribed by a doctor OR currently on a daily beta-blocker or statin regimen prescribed by a doctor
8. Some comfort using technology such as electronic tablets or smartphones

Exclusion Criteria:

1. Deemed unable to comply with the protocol (either self-selected or by indicating during screening that s/he could not complete all requested tasks). This includes patients with a level of cognitive impairment indicative of dementia and patients with current alcohol or substance abuse;
2. Deemed to need immediate psychiatric intervention (that is, has to be hospitalized or have some other psychiatric intervention within 72 hours);
3. Unavailable for follow-up. This includes patients with a terminal noncardiovascular illness (life expectancy less than 1 year by physician report) and those who indicate they are about to leave the United States;
4. Underwent a surgical procedure within the past 24 hours and/or is scheduled for a surgical procedure within the next 24 hours.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2019-03-28 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey L Birk, PhD, Principal Investigator — Columbia University
Locations (1):
- NewYork-Presbyterian/Columbia University Irving Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lopez-Veneros D, Cumella R, Kronish IM, Lazarov A, Birk JL. Home-based cognitive bias modification training for reducing maladaptive fear in patients with suspected acute coronary syndrome: a pilot randomized clinical trial. Pilot Feasibility Stud. 2024 Jan 11;10(1):7. doi: 10.1186/s40814-024-01442-2. PMID 38212853
- [Derived] Birk JL, Cumella R, Lopez-Veneros D, Jurado A, Romero EK, Lazarov A, Kronish IM. Intervening on fear after acute cardiac events: Rationale and design of the INFORM randomized clinical trial. Health Psychol. 2020 Sep;39(9):736-744. doi: 10.1037/hea0000853. PMID 32833475

RESULTS

PARTICIPANT FLOW:
Recruitment Details: English and Spanish-speaking patients with Elevated Threat Perception Scores were recruited for enrollment from a parent study after a suspected Acute Coronary Syndrome (ACS) event. Patients were recruited both in hospital (on cardiac floors), as well as at home or in-clinic after discharge.
Pre-assignment Details: Twenty-six patients consented to the study. After consent, all participants were asked to complete a baseline questionnaire and a brief training with a demo tablet. Two participants decided to withdraw from the study, and four participants were administratively withdrawn by the PI as they were determined to be unable to comply with protocol (e.g., unable to complete tablet demo) and therefore not eligible for the study. These six participants were not assigned study groups.
Period: Overall Study
Arm/Group | Cognitive Bias Modification Training | Attention Control Training
Started | 11 | 9
Completed | 10 | 7
Not Completed | 1 | 2
Not completed — Extenuating Circumstances (COVID-19 pandemic) | 1 | 0
Not completed — Other (e.g., too busy) | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cognitive Bias Modification Training | Attention Control Training | Total
Number analyzed (Participants) | 11 | 9 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.00 (13.20) | 59.88 (13.69) | 60.00 (13.20)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Sex: Male | 5 | 5 | 10
  Sex: Female | 6 | 4 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 4 | 10
  Not Hispanic or Latino | 5 | 5 | 10
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 1 | 4
  White | 2 | 3 | 5
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 6 | 5 | 11
Region of Enrollment [Number; unit: participants]
  United States | 11 | 9 | 20

OUTCOME MEASURES:

1. Primary Outcome: Change in Total Score for Concerns About Recurrence Scale [Adapted for Acute Coronary Syndrome]
Description: This 19-item self-report scale measures fear of recurrence of ACS events. It uses a 5-point Likert scale (0 to 4). It has three subscales: health worries (items 1-11; subscale range: 0-44), role worries (items 12-17: subscale range: 0-24), and death worries (items 18-19: subscale range: 0-8). The total score is computed as the sum of all items in the scale (total score range: 0 to 76). Higher total scores indicate greater fear of recurrence. The study will test whether there is a larger Time-1-to-Time-2 reduction in Concerns about Recurrence total scores for the intervention group relative to the control group. The outcome for each group is computed as mean of the difference of the Time-2 score minus the Time-1 score. This is the sole primary outcome because the trial design was statistically powered to reduce FoR.
Time Frame: Pre-Training/Time 1, Post-Training/Time 2 (approximately 4 weeks apart)
Population: The number of participants analyzed is the number of participants who completed Visit 1 and Visit 2 such that the change score outcome could be computed. Only the subjects that completed both visits were included in the analysis (10 out of 11 subjects in intervention group and 7 out of 9 subjects in placebo group).
Measure: Mean (Standard Deviation); unit: change in score on a scale
Arm/Group | Cognitive Bias Modification Training | Attention Control Training
Number analyzed (Participants) | 10 | 7
change in score on a scale | -5.40 (19.55) | -2.86 (3.93)
Statistical Analysis 1: Comparison: Cognitive Bias Modification Training vs Attention Control Training; Test type: Superiority; p = 0.698, t-test, 2 sided; The p-value is adjusted using the Satterthwaite correction due to unequal variances between the two groups; Mean difference (in change score) = 2.54, 95% CI 2-sided [-11.62 to 16.71] — A higher value of the estimation parameter of mean difference in change score indicates a greater reduction in the measure for the intervention group relative to the attention control group

2. Secondary Outcome: Total Score for Self-reported Extent of Nonadherence to Medication From the Extent of and Reasons for Nonadherence Scale [Adapted]
Description: The self-reported scale called the Extent of and Reasons for Nonadherence Scale [Adapted] measures how often participants do not take their prescribed medication and the reasons that they were nonadherent (e.g., forgot, out of routine, feeling down or upset). The measure of extent of nonadherence is the total of 3 items in the extent portion of the scale such that higher scores represent greater nonadherence (total score range: 3-15). The study will test whether there are lower self-reported extent of nonadherence scores for the intervention group relative to the control group at time 2. (Because not all participants are expected at time 1 to have been already taking the particular heart medication assessed in the study, the self-reported questions about medication adherence are only administered at time 2.)
Time Frame: Post-Training/Time 2 (approximately 4 weeks after Time 1)
Population: The number of participants analyzed is the number of participants who completed Visit 2 such that the outcome score could be computed. Only the subjects that completed this questionnaire at Visit 2 were included in the analysis (7 out of 11 subjects in intervention group and 6 out of 9 subjects in placebo group).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cognitive Bias Modification Training | Attention Control Training
Number analyzed (Participants) | 7 | 6
score on a scale | 11.71 (4.39) | 7.83 (3.92)
Statistical Analysis 1: Comparison: Cognitive Bias Modification Training vs Attention Control Training; Note that the measure of extent of medication nonadherence used the older 5-item version of the scale rather than the newer 3-item version of the scale because the IRB modification to change the measure took effect after the majority of participants who provided data for Visit 2 had completed the measure; Test type: Superiority; p = 0.123, t-test, 2 sided; Mean Difference (Final Values) = -3.88, 95% CI 2-sided [-9.00 to 1.24] — A lower value of the estimation parameter of mean difference indicates lower extent of medication nonadherence for the intervention relative to the control group

3. Secondary Outcome: Change in Total Score for the International Physical Activity Questionnaire in MET Minutes/Week
Description: This 7-item self-report scale measures the extent to which participants engaged in physical activity at a variety of intensity levels during the last week. Higher scores represent greater total metabolic equivalent of task (MET) minutes of physical activity per week based on the following estimates: 3.3 MET units for walking, 4.4 MET units for moderate activity, 8 MET units for vigorous activity. The study will test whether there is a larger Time-1-to-Time-2 increase in total scores on the International Physical Activity Questionnaire (units: MET minutes/week) for the intervention group relative to the control group. The outcome for each group is computed as mean of the difference of the Time-2 score minus the Time-1 score.
Time Frame: Pre-Training/Time 1, Post-Training/Time 2 (approximately 4 weeks apart)
Population: The number of participants analyzed is the number of participants who completed Visit 1 and Visit 2 such that the change score outcome could be computed. Only the subjects that completed this questionnaire at both visits were included in the analysis (9 out of 11 subjects in intervention group and 7 out of 9 subjects in placebo group).
Measure: Mean (Standard Deviation); unit: change in MET minutes/week
Arm/Group | Cognitive Bias Modification Training | Attention Control Training
Number analyzed (Participants) | 9 | 7
change in MET minutes/week | 648.3 (3039.3) | 714.6 (2734.2)
Statistical Analysis 1: Comparison: Cognitive Bias Modification Training vs Attention Control Training; Test type: Superiority; p = 0.965, t-test, 2 sided; Mean difference (in change score) = 66.29, 95% CI 2-sided [-3081.7 to 3214.3]

4. Secondary Outcome: Change in Cue Presence Score for the Context Sensitivity Index
Description: This self-report scale measures participants' ability to identify information about stressful situations that may be helpful for successfully and flexibly regulating unpleasant feelings of distress. In particular, the cue presence score reflects the sensitivity to the presence of meaningful contextual cues. This cue presence score is calculated as the sum of 10 relevant items from the scale. Greater cue presence scores indicate greater context sensitivity (cue presence score range: 10-77). The study will test whether there is a larger Time-1-to-Time-2 increase in cue presence scores on the Context Sensitivity Index for the intervention group relative to the control group. The outcome for each group is computed as mean of the difference of the Time-2 score minus the Time-1 score.
Time Frame: Pre-Training/Time 1, Post-Training/Time 2 (approximately 4 weeks apart)
Population: The number of participants analyzed is the number of participants who completed Visit 1 and Visit 2 such that the change score outcome could be computed. Only the subjects that completed this questionnaire at both visit were included in the analysis (10 out of 11 subjects in intervention group and 7 out of 9 subjects in placebo group).
Measure: Mean (Standard Deviation); unit: change in score on a scale
Arm/Group | Cognitive Bias Modification Training | Attention Control Training
Number analyzed (Participants) | 10 | 7
change in score on a scale | 0.60 (12.59) | -5.57 (9.36)
Statistical Analysis 1: Comparison: Cognitive Bias Modification Training vs Attention Control Training; Test type: Superiority; p = 0.290, t-test, 2 sided; Mean difference (in change score) = -6.17, 95% CI 2-sided [-18.15 to 5.81] — A higher value of the estimation parameter of mean difference in change score indicates a greater increase in context sensitivity for the intervention group relative to the attention control group

5. Secondary Outcome: Change in Total Score for Future Time Perspective Scale
Description: This 10-item self-reported scale measures participants' perceptions of their own futures as either limited (lower scores) or expansive (higher scores). The total score is the sum of all 10 items after three of the items (8-10) have been reverse-coded (total score range: 10-77). The study will test whether there is a larger Time-1-to-Time-2 increase in Future Time Perspective total scores for the intervention group relative to the control group. The outcome for each group is computed as mean of the difference of the Time-2 score minus the Time-1 score.
Time Frame: Pre-Training/Time 1, Post-Training/Time 2 (approximately 4 weeks apart)
Population: Only the subjects that completed this questionnaire at both visit were included in the analysis (10 out of 11 subjects in intervention group and 7 out of 9 subjects in placebo group).
Measure: Mean (Standard Deviation); unit: change in score on a scale
Arm/Group | Cognitive Bias Modification Training | Attention Control Training
Number analyzed (Participants) | 10 | 7
change in score on a scale | 2.30 (11.84) | -2.77 (14.12)
Statistical Analysis 1: Comparison: Cognitive Bias Modification Training vs Attention Control Training; Test type: Superiority; p = 0.434, t-test, 2 sided; Mean difference (in change score) = -5.07, 95% CI 2-sided [-18.51 to 8.38] — A higher value of the estimation parameter of mean difference in change score indicates a greater increase in future time perspective for the intervention group relative to the attention control group

6. Secondary Outcome: Percentage of Adherent Days to Medication (Aspirin, Beta-blocker, or Statin)
Description: Participants' post-hospitalization medication adherence is measured objectively through electronically recorded pill bottle openings using the eCAP device (Information Mediary Corp., Ottawa, Canada). The measure is operationalized as the percentage of adherent days. The study will test whether there is a higher percentage of adherent days across the entire study monitoring period for the intervention group relative to the control group.
Time Frame: Up to 2 months (starting after Pre-Training/Time 1 and extending for approximately 4 weeks after Post-Training/Time 2)
Population: Only the subjects that used the eCAP device to monitor their heart medication adherence were included in the analysis (9 out of 11 subjects in intervention group and 6 out of 9 subjects in placebo group).
Measure: Mean (Standard Deviation); unit: percentage of days
Arm/Group | Cognitive Bias Modification Training | Attention Control Training
Number analyzed (Participants) | 9 | 6
percentage of days | 61.78 (35.38) | 78.83 (24.77)
Statistical Analysis 1: Comparison: Cognitive Bias Modification Training vs Attention Control Training; Test type: Superiority; p = 0.293, t-test, 2 sided; Mean Difference (Final Values) = 17.05, 95% CI 2-sided [-19.07 to 53.17] — A higher value of the estimation parameter of mean difference indicates a lower extent of objectively measured medication adherence for the intervention relative to the control group

ADVERSE EVENTS:
Time Frame: Adverse event data were assessed during the time period in which participants engaged in study procedures from the time of enrollment until the time of the final study visit (i.e., approximately 5 weeks).
Arm/Group | Cognitive Bias Modification Training | Attention Control Training
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/9
Other Adverse Events (participants affected / at risk) | 0/11 | 0/9

LIMITATIONS AND CAVEATS:
Because New York City was the original epicenter of the COVID-19 outbreak in the US, the pandemic brought study enrollment to a halt in March 2020. Our potential pool of participants from the parent study also slowed due to the implementation of a new test (high sensitivity cardiac troponin assay) to diagnose ACS in the emergency department. Although beneficial for patient treatment, it reduced the number of patients enrolled in the parent study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-06-21): https://cdn.clinicaltrials.gov/large-docs/13/NCT03853213/Prot_SAP_000.pdf